CLINICAL TRIAL: NCT06932627
Title: Effects of Intravascular Laser Irradiation of Blood for Mitochondral Dysfunction and Oxidative Stress in Adults With Chronic Cerebral Ischemic Stroke
Brief Title: Effects of Intravascular Laser Irradiation of Blood for Mitochondral Dysfunction in Cerebral Ischemic Stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tri-Service General Hospital (Other)
Responsible Party: Principal Investigator, Liang-Cheng Chen, Attending Physician and lecturer of Department of Physical Medicine and Rehabilitation, Tri-Service General Hospital
Allocation: Not Applicable | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TSGH-D-111109
Record Dates: First submitted 2025-04-10; First posted 2025-04-17 (Actual); Last update posted 2025-04-17 (Actual); Status verified 2024-04

CONDITIONS: Ischemic Stroke
Keywords: Ischemic Stroke; intravenous laser irradiation of blood; mitochondria activity
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ILIB therapy (Experimental): The treatment group receive an intravenous helium-neon laser phototherapy. A vein indwelling needle will be placed in their veins located in the upper elbow, and the laser fiber catheter will be introduced through the indwelling cannula. The laser power is set between 5 Mw, 30 minutes each time, once everyother day for 3 consecutive days each week, for 2 weeks (total 6 times in one course)
  Interventions: Procedure: ILIB
- sham control (Sham Comparator): The steps for the control group are the same as the treatment group, except that the output power is adjusted to zero intensity.
  Interventions: Procedure: Sham Control

INTERVENTIONS:
Procedure: ILIB — The treatment group receive an intravenous laser phototherapy. A vein indwelling needle will be placed in their veins located in the upper elbow, and the laser fiber catheter will be introduced through the indwelling cannula. The laser power is set between 5 Mw, 30 minutes each time,once every other day for 3 consecutive days each week, for 2 weeks (total 6 times in one course)
  Arms: ILIB therapy
Procedure: Sham Control — The steps for the control group are the same as the treatment group, exceptthat the output power is adjusted to zero intensity.
  Arms: sham control

SUMMARY:
Background : This research is designed through randomization, control, and double-blind trial to explore the clinical effectiveness of intravenous laser irradiation of blood for ischemic stroke patient; The research will further explore the changes of mitochondria function after treatment. The light accelerates blood and cells circulation in the human body, so that protein molecular structure would promote changes. Pain control is indicated in such treatment, but still lacking evidence of neurological symptoms and functional improvement.

Purpose:This research is designed through randomization, control, and double-blind trial to therapeutic effect and platelet activity after intravenous laser irradiation of blood for ischemic stroke patient. Furthermore, to establish a new way of clinical therapy.

Method: The investigators plan to recruit 20 patients who are between the ages of 20 to 80 years old. The participants are required to have clear conscious and be able to communicate. The patient with mild to moderate stroke ( NIHSS=1-15), which onset between one month to 2 years will be included. The treatment group will receive an intravenous helium-neon laser phototherapy. A vein indwelling needle will be placed in their veins located in the upper elbow, and the laser fiber catheter will be introduced through the indwelling cannula. The power is set between 5Mw, 30 minutes each time, once everyother day for 3 days each week, for 2 weeks (total 6 times in one course). The steps for the control group are the same, except that the output power is adjusted to zero intensity. This plan will be explained to the patient in detail during the outpatient visit and patients will sign the consent form upon agreement. Before intravenous laser irradiation,three days, one month, and three months after the therapy, 20 ml of autologous peripheralvenous blood need to be drawn for basic blood tests and platelet activity tests. At the same time, the clinical functions of patients will be evaluated, including NIHSS, mRS.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 20 to 80 years old
* Able to speak and understand Mandarin/Taiwanese
* No cognitive impairment
* Residual motor function impairment (mRS>1)
* Mild stroke (NIHSS=1-4) or Moderate stroke(NIHSS=5-15)
* No psychological disease

Exclusion Criteria:

* Severe stroke (NIHSS=16-42)
* History of intracerebral hemorrhage and other major surgery
* History of malignancy, chronic kidney disease
* Active infection
* Chronic hepatitis B or Chronic hepatitis C
* Unstable angina or acute myocardial infarction within 6 months
* Severe cognition impairment
* Pregnancy

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2023-08-01 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
National Institutes of Health Stroke Scale (NIHSS) | 3 month
  NIHSS is a measure of the severity of symptoms associated with ischemic strokeand is used as a quantitative measure of neurological deficit post stroke. NIHSSscore is composed of 11 items, including consciousness, eye movement, visualfields, muscle power of four limbs, limbs ataxia, sensation, language, dysarthria andextinction. Each of which scores a specific ability between a 0 and 4. For each item,a score of 0 typically indicates normal function in that specific ability, while a higherscore is indicative of some level of impairment. Total score are between 0-42.
  Measure before intravenous laser irradiation, three days, one month, and threemonths after the therapy.

SECONDARY OUTCOMES:
Modified Rankin Scale (mRS) | 3 month
  The Modified Rankin Scale (mRS) is used to measure the degree of disability ordependence in the daily activities in patients who have had a stroke 0: Nosymptoms at all

CONTACTS AND LOCATIONS:
Locations (1):
- Tri-service general hospital, Taipei, Taiwan